CLINICAL TRIAL: NCT03400943
Title: A Randomized, Parallel-group, Double-blind and Open-label Placebo-controlled, Multicenter Study to Assess the Efficacy and Safety of Vilaprisan in Subjects With Uterine Fibroids
Brief Title: Assess Safety and Efficacy of Vilaprisan in Subjects With Uterine Fibroids (ASTEROID 3)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to a change in the development program, the study was closed prematurely.
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 15787; 2017-002997-38 (EudraCT Number)
Record Dates: First submitted 2018-01-05; First posted 2018-01-17 (Actual); Results first posted 2021-06-11 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Uterine Fibroids
Keywords: Heavy menstrual bleeding
MeSH Terms: conditions — Leiomyoma; Menorrhagia | interventions — vilaprisan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Blinding will be applied to Treatment Groups A1, B1, and B2; Treatment Group A2 will be open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Vilaprisan (A1) (Experimental): Vilaprisan (2 mg) in treatment period 1 for 12 weeks and in treatment period 2 for 12 weeks, separated by 1 bleeding episode.
  Interventions: Drug: Vilaprisan (BAY1002670); Drug: Placebo
- Vilaprisan (A2) (Experimental): Vilaprisan (2 mg) in treatment period 1 for 12 weeks and in treatment period 2 for 12 weeks without a break.
  Interventions: Drug: Vilaprisan (BAY1002670)
- Placebo+Vilaprisan (B1) (Experimental): Placebo in treatment period 1 for 12 weeks, and vilaprisan (2 mg) in treatment period 2 for 12 weeks, separated by 1 bleeding episode.
  Interventions: Drug: Vilaprisan (BAY1002670); Drug: Placebo
- Vilaprisan+Placebo (B2) (Experimental): Vilaprisan (2 mg) in treatment period 1 for 12 weeks and placebo in treatment period 2 for 12 weeks, separated by 1 bleeding episode.
  Interventions: Drug: Vilaprisan (BAY1002670); Drug: Placebo

INTERVENTIONS:
Drug: Vilaprisan (BAY1002670) — 2 mg of Vilaprisan once daily up to 2 x 12 weeks
Drug: Placebo — Matching placebo was administered to group B1 and B2.
  Arms: Placebo+Vilaprisan (B1); Vilaprisan (A1); Vilaprisan+Placebo (B2)

SUMMARY:
The primary objective of this study was to show superiority in the treatment of HMB of vilaprisan in subjects with uterine fibroids compared to placebo.

The secondary objectives of this study were to additionally evaluate the efficacy and safety of vilaprisan in subjects with uterine fibroids.

ELIGIBILITY:
Inclusion Criteria:

* Women, 18 years or older in good General health
* Diagnosis of uterine fibroid(s) documented by ultrasound at screening with at least 1 fibroid with largest Diameter ≥ 30 mm and < 120 mm
* Heavy menstrual bleeding (HMB) in at least 2 bleeding periods during the Screening period each with blood loss volume of >80.00 mL documented by alkaline hematin (AH) method
* An endometrial biopsy performed during the Screening period without significant histological disorder such as endometrial hyperplasia (including simple hyperplasia) or other significant endometrial pathology
* Use of an acceptable non-hormonal method of contraception (ie, either male condom, cap, diaphragm or sponge, each in combination with spermicide) starting at Visit 1 until the end of the study

Exclusion Criteria:

* Pregnancy or lactation (less than 3 month since delivery, abortion, or lactation before start of Treatment)
* Hypersensitivity to any ingredient of the study drug
* Any condition requiring immediate blood transfusion
* Laboratory values outside inclusion range before randomization and considered as clinically relevant.
* Any diseases, conditions, or medications that can compromise the function of the body systems and could result in altered absorption, excessive accumulation, impaired metabolism, or altered excretion of the study drug
* Any diseases or conditions that might interfere with the conduct of the study or the interpretation of the results
* Abuse of alcohol, drugs, or medicines (eg, laxatives)
* Use of other treatments that might interfere with the conduct of the study or the interpretation of the results
* Undiagnosed abnormal genital bleeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2018-01-17 (Actual); Primary Completion 2019-06-09 (Actual); Study Completion 2022-04-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (103):
- United States (52):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - California Center for Clinical Research, Arcadia, California
  - Core Healthcare Group, Cerritos, California
  - AVIVA Research, Escondido, California
  - National Research Institute - Los Angeles, Los Angeles, California
  - Harbor - UCLA Medical Center, Torrance, California
  - Ideal Clinical Research, Aventura, Florida
  - South Florida Medical Research, Aventura, Florida
  - Helix Biomedics, LLC, Boynton Beach, Florida
  - Dr. Victoria Garcia & Associates, LLC Doral Medical Research, Doral, Florida
  - Sweet Hope Research Specialty, Inc. - Hialeah, Hialeah, Florida
  - Clinical Neurosciences Solutions, Inc. DBA CNS Healthcare, Jacksonville, Florida
  - Altus Research, Lake Worth, Florida
  - Axcess Medical Research, LLC, Loxahatchee Groves, Florida
  - Ocean Blue Medical Research Center, Inc., Miami Springs, Florida
  - Accelerated Enrollment Solutions a business of PPD, Orlando, Florida
  - Discovery Clinical Research, Plantation, Florida
  - ONCOVA Clinical Research, Inc., Saint Cloud, Florida
  - Georgia Center For Women, Atlanta, Georgia
  - Agile Clinical Research Trials, LLC, Atlanta, Georgia
  - Atlanta Women's Research Institute, Inc. - Alpharetta, Atlanta, Georgia
  - Medisense, Inc., Atlanta, Georgia
  - Paramount Research Solutions-College Park, College Park, Georgia
  - One Health Research Clinic, Norcross, Georgia
  - Fellows Research Alliance - Savannah, Savannah, Georgia
  - GTC Research, Shawnee Mission, Kansas
  - Omni Fertility and Laser Institute, Shreveport, Louisiana
  - PharmaSite Research, Inc., Baltimore, Maryland
  - Simmonds, Martin and Helmbrecht, Gaithersburg, Maryland
  - Advantia Health, LLC Obstetrics & Gynecology Assoc., Silver Spring, Maryland
  - SUNY Downstate Medical Center, Brooklyn, New York
  - Carolinas Healthcare System, Charlotte, North Carolina
  - Unified Women's Clinical Research - Morehead City, Morehead City, North Carolina
  - Eastern Carolina Women's Center, New Bern, North Carolina
  - Wake Research, Inc., Raleigh, North Carolina
  - Main Line Fertility Center, Bryn Mawr, Pennsylvania
  - Clinical Research of Philadelphia, LLC, Philadelphia, Pennsylvania
  - Fellows Research Alliance, Inc., Bluffton, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Fusion Clinical Research of Spartanburg, LLC, Spartanburg, South Carolina
  - Chattanooga Medical Research, LLC, Chattanooga, Tennessee
  - Clinical Neurosciences Solutions, Inc DBA CNS Healthcare, Memphis, Tennessee
  - Paramount Research Solutions-Nashville, Nashville, Tennessee
  - Texas Health Care, PLLC, Fort Worth, Texas
  - Willowbend Health & Wellness Associates, Frisco, Texas
  - Family Medicine Clinic, Georgetown, Texas
  - Biopharma Informatic, Inc., Houston, Texas
  - Centex Studies, Inc., Houston, Texas
  - The Center for Clinical Trials, Inc., Houston, Texas
  - Houston Center for Clinical Research, LLC, Sugar Land, Texas
  - Millennium Clinical Trials, LLC, Arlington, Virginia
  - Synexus Research, LLC, Richmond, Virginia
- Bulgaria (4):
  - Multiprofile Hospital for Active Treatment-Dr. T. Venkova AD, Gabrovo
  - Hospital for Active Treatment - Prof.Paraskev Stoyanov AD, Lovech
  - MHAT Dr. Bratan Shukerov AD, Smolyan
  - MHAT for Women's Health - Nadezhda OOD, Sofia
- China (29):
  - 900th Hospital of Joint Logistics Support Force, Fuzhou, Fujian
  - Guangzhou Women and Children's Medical Center, Guangzhou, Guangdong
  - The Third Affiliated Hospital, Sun Yat-Sen University, Guangzhou, Guangdong
  - Boai Hospital of Zhongshan, Zhongshan, Guangdong
  - Hainan General Hospital, Haikou, Hainan
  - Wuhan Tongji Reproductive Medicine Hospital, Wuhan, Hubei
  - Nanjing Maternity and Child Health Care Hospital, Nanjing, Jiangsu
  - NJ Drum Tower Hospital, the Affil Hos of NJ Univ Med School, Nanjing, Jiangsu
  - Zhongda Hospital Southeast University, Nanjing, Jiangsu
  - 1st Affiliated hospital of Soochow University, Suzhou, Jiangsu
  - Jiangxi Maternal and Child Health Hospital, Nanchang, Jiangxi
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - The First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - The Second Affiliated Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - Women's Hospital School of Medicine Zhejiang University, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital, Zhejiang University School of Med, Hangzhou, Zhejiang
  - The Second Affliated Hospital of Wenzhou Medicial University, Wenzhou, Zhejiang
  - Beijing Hospital of Traditional Chinese Medicine, Beijing
  - Peking University First Hospital, Beijing
  - Beijing Friendship Hospital, Capital Medical University, Beijing
  - Beijing Tiantan Hospital, Captial Medical University, Beijing
  - Shanghai East Hospital Affiated to Tongji University, Shanghai
  - Tianjin Medical University General Hospital, Tianjin
- Czechia (4):
  - Gynekologie MEDA s.r.o., Brno
  - Soukroma gynekologicka ambulance, Fulnek
  - Gynekologie Studentsky dum s.r.o., Prague
  - MUDr. Ivana Salamonova s.r.o., Vysoké Mýto
- Israel (4):
  - Clalit Health Services through HaEmek Medical Center, Afula
  - Hillel Yaffe Medical Center, Hadera
  - Lady Davis Carmel Medical Center, Haifa
  - Meir Medical Center, Kfar Saba
- Malaysia (3):
  - University Hospital Kebangsaan Malaysia, Kuala Lumpur
  - Hospital Wanita dan Kanak-Kanak Sabah, Sabak Bernam
  - Sarawak General Hospital, Sarawak
- New Zealand (2):
  - P3 Research Ltd Hawkes Bay, Hawkes Bay
  - P3 Research, Tauranga
- KK Women's and Children's Hospital, Singapore, Singapore
- South Africa (4):
  - Dr L Reynders Practice, Lyttelton Manor, Gauteng
  - Wilgeheuwel Hospital, Roodepoort, Gauteng
  - Umhlanga Medical Centre, Durban, KwaZulu-Natal
  - Ethekwini Hospital & Heart Centre, Durban, KwaZulu-Natal

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- [Derived] Al-Hendy A, Zhou YF, Faustmann T, Groettrup-Wolfers E, Laapas K, Parke S, Seitz C. Efficacy and safety of vilaprisan in women with uterine fibroids: data from the ASTEROID 3 randomized controlled trial. F S Sci. 2023 Nov;4(4):317-326. doi: 10.1016/j.xfss.2023.06.003. Epub 2023 Jul 10. PMID 37437885
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 104 study centers in 9 countries worldwide between 17-Jan-2018 (first participant first visit) and 06-Apr- 2022 (last participant last visit).
Pre-assignment Details: Overall, 646 participants were screened. Of the 646 screened participants, 553 (85.6%) participants were not randomized to treatment. The majority of these (n=403) were screen failures. Of the 93 participants who were randomized, 79 participants received study treatment.
Period: Treatment Period 1
Arm/Group | Vilaprisan (A1) | Vilaprisan (A2) | Placebo+Vilaprisan (B1) | Vilaprisan+Placebo (B2)
Started (Randomized) | 23 | 23 | 24 | 23
Treated | 18 | 21 | 20 | 20
Completed | 18 | 21 | 18 | 18
Not Completed | 5 | 2 | 6 | 5
Not completed — Adverse Event | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 1 | 0
Not completed — Study terminated by sponsor | 2 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 3 | 1
Not completed — Other | 2 | 1 | 2 | 2
Period: Post-treatment Period 1
Arm/Group | Vilaprisan (A1) | Vilaprisan (A2) | Placebo+Vilaprisan (B1) | Vilaprisan+Placebo (B2)
Started | 18 | 0 | 18 | 18
Completed | 7 | 0 | 7 | 5
Not Completed | 11 | 0 | 11 | 13
Not completed — Adverse Event | 2 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0
Not completed — Study terminated by sponsor | 5 | 0 | 5 | 6
Not completed — Withdrawal by Subject | 1 | 0 | 2 | 2
Not completed — Other | 2 | 0 | 4 | 5
Period: Treatment Period 2
Arm/Group | Vilaprisan (A1) | Vilaprisan (A2) | Placebo+Vilaprisan (B1) | Vilaprisan+Placebo (B2)
Started (Treatment started) | 7 | 21 | 7 | 5
Completed | 6 | 13 | 7 | 5
Not Completed | 1 | 8 | 0 | 0
Not completed — Study terminated by sponsor | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Not completed — Other | 1 | 6 | 0 | 0
Period: Follow-up Period
Arm/Group | Vilaprisan (A1) | Vilaprisan (A2) | Placebo+Vilaprisan (B1) | Vilaprisan+Placebo (B2)
Started | 7 | 15 | 7 | 5
Completed | 6 | 15 | 7 | 5
Not Completed | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: SAF consisted of all randomized participants in FAS who took at least 1 dose of study drug. The discrepancy of group B1 and B2 between subject dispostion and baseline characteristics was caused by mistakes in the administration of study drug.
  Three participants who were assigned to B1, erroneously received vilaprisan treatment instead of placebo in Treatment Period (TP) 1. Two participants who were assigned to B1, erroneously received placebo instead of vilaprisan in TP2.
Groups:
- Total: Total of all reporting groups
Arm/Group | Vilaprisan (A1) | Vilaprisan (A2) | Placebo+Vilaprisan (B1) | Vilaprisan+Placebo (B2) | Total
Number analyzed (Participants) | 18 | 21 | 17 | 23 | 79
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.1 (4.4) | 43.1 (5.8) | 42.5 (5.3) | 43.8 (5.1) | 43.2 (5.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 21 | 17 | 23 | 79
  Male | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 1 | 1 | 0 | 6
  Not Hispanic or Latino | 13 | 20 | 16 | 22 | 71
  Unknown or Not Reported | 1 | 0 | 0 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 5 | 8 | 5 | 7 | 25
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 6 | 5 | 7 | 11 | 29
  White | 7 | 6 | 5 | 5 | 23
  More than one race | 0 | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1
Endometrial thickness [Mean (Standard Deviation); unit: Millimeters] — Ultrasound examinations were performed. Endometrial thickness was measured in the medio-sagittal section as double-layer in millimeters. Baseline data of endometrial thickness is provided in the table. Population: Participants in safety analysis set (SAF) with endometrial thickness measured and analyzed.
  Millimeters
    number analyzed (Participants) | 18 | 20 | 17 | 22 | 77
    (all) | 13.6 (7.6) | 11.0 (5.4) | 11.9 (6.5) | 10.5 (3.9) | 11.7 (5.9)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Amenorrhea
Description: Amenorrhea was defined as menstrual blood loss (MBL) <2 mL during the last 28 days of treatment measured by the alkaline hematin (AH) method.
Time Frame: The last 28 days of treatment period 1
Population: FAS was analysed. FAS consists of all randomized participants, excluding randomized participants who did not start treatment period 1 due to the study being temporarily on hold, including 84 participants. Participants were analyzed as randomized.
Measure: Count of Participants; unit: Participants
Arm/Group | Vilaprisan (A1) | Vilaprisan (A2) | Placebo+Vilaprisan (B1) | Vilaprisan+Placebo (B2)
Number analyzed (Participants) | 20 | 23 | 20 | 21
Participants | 16 | 20 | 4 | 15
Statistical Analysis 1: Comparison: Vilaprisan (A1) vs Placebo+Vilaprisan (B1) vs Vilaprisan+Placebo (B2); Vilaprisan (A1) and Vilaprisan+Placebo (B2) combined vs. Placebo+Vilaprisan (B1) in treatment period 1; Test type: Superiority; p < .0001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 0.56, 95% CI 2-sided [0.33 to 0.78] — Number of subjects per treatment: 41 (Vilaprisan) / 20 (Placebo)

2. Secondary Outcome: Number of Participants With Heavy Menstrual Bleeding (HMB) Response
Description: HMB response was defined as MBL <80 mL during the last 28 days of treatment and >50% reduction from baseline based on AH-method.
Time Frame: The last 28 days of treatment period 1 and treatment period 2
Population: FAS population was analysed.
Measure: Count of Participants; unit: Participants
Arm/Group | Vilaprisan (A1) | Vilaprisan (A2) | Placebo+Vilaprisan (B1) | Vilaprisan+Placebo (B2)
Number analyzed (Participants) | 20 | 23 | 20 | 21
Participants
  Treatment period 1 | 17 | 20 | 8 | 17
  Treatment period 2: number analyzed (Participants) | 7 | 15 | 7 | 5
  Treatment period 2 | 6 | 14 | 6 | 1

3. Secondary Outcome: Time to Onset of Amenorrhea
Description: Onset of amenorrhea was defined by the first day for which the MBL for all subsequent 28-day periods up to the end of a treatment period was < 2 mL (amenorrhea defined similar to primary endpoint).
Time Frame: In treatment period 1 (12 weeks) and in treatment period 2 (12 weeks)
Population: FAS population was analysed. In treatment period 2, participants who did not start the respective treatment period or had less than 28 days of treatment are included among censored observations.
  For treatment arm Vilaprisan (A2), the combined data of treatment period 1 and treatment period 2 were entered.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Vilaprisan (A1) | Vilaprisan (A2) | Placebo+Vilaprisan (B1) | Vilaprisan+Placebo (B2)
Number analyzed (Participants) | 20 | 23 | 20 | 21
Days
  Treatment Period 1 | 3 [2 to 4] | NA [NA to NA] — NA: not applicable. For treatment arm Vilaprisan (A2), the combined data of treatment period 1 and treatment period 2 were entered. | NA [NA to NA] — NA indicates that the value cannot be estimated due to censored data. | 6 [1 to 46]
  Treatment Period 2 | 21 [2 to 32] | NA [NA to NA] — NA: not applicable. For treatment arm Vilaprisan (A2), the combined data of treatment period 1 and treatment period 2 were entered. | 2 [1 to NA] — NA indicates that the value cannot be estimated due to censored data. | NA [NA to NA] — NA indicates that the value cannot be estimated due to censored data.
  Treatment periods 1 and 2 combined | NA [NA to NA] — NA: not applicable. | 9 [3 to 107] | NA [NA to NA] — NA: not applicable. | NA [NA to NA] — NA: not applicable.

4. Secondary Outcome: Time to Onset of Controlled Bleeding
Description: Onset of controlled bleeding was defined by the first day for which the MBL for all subsequent 28-day periods up to the end of a treatment period was <80.00 mL based on AH-method.
Time Frame: In treatment period 1 (12 weeks) and in treatment period 2 (12 weeks)
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Vilaprisan (A1) | Vilaprisan (A2) | Placebo+Vilaprisan (B1) | Vilaprisan+Placebo (B2)
Number analyzed (Participants) | 20 | 23 | 20 | 21
Days
  Treatment period 1 | 1 [1 to 2] | NA [NA to NA] — NA: not applicable. For treatment arm Vilaprisan (A2), the combined data of treatment period 1 and treatment period 2 were entered. | NA [53 to NA] — NA indicates that the value cannot be estimated due to censored data. | 1 [1 to 1]
  Treatment period 2 | 1 [1 to 1] | NA [NA to NA] — NA: not applicable. For treatment arm Vilaprisan (A2), the combined data of treatment period 1 and treatment period 2 were entered. | 1 [1 to 2] | NA [NA to NA] — NA indicates that the value cannot be estimated due to censored data.
  Treatment periods 1 and 2 combined | NA [NA to NA] — NA: not applicable. | 1 [1 to 7] | NA [NA to NA] — NA: not applicable. | NA [NA to NA] — NA: not applicable.

5. Secondary Outcome: Number of Participants With Absence of Bleeding (Spotting Allowed)
Description: Absence of bleeding was defined as no scheduled or unscheduled bleeding (spotting allowed) during the last 28 days of a treatment period based on subjects' daily responses to the Uterine Fibroid Daily Bleeding Diary (UF-DBD).
Time Frame: The last 28 days of treatment period 1 and treatment period 2
Population: FAS population was analysed.
Measure: Count of Participants; unit: Participants
Arm/Group | Vilaprisan (A1) | Vilaprisan (A2) | Placebo+Vilaprisan (B1) | Vilaprisan+Placebo (B2)
Number analyzed (Participants) | 20 | 23 | 20 | 21
Participants
  Treatment period 1 | 16 | 20 | 4 | 15
  Treatment period 2: number analyzed (Participants) | 7 | 15 | 7 | 5
  Treatment period 2 | 6 | 13 | 6 | 0

6. Secondary Outcome: Number of Participants With Endometrial Histology Findings by Endometrial Biopsy Main Results (Majority Read, Main Diagnosis)
Description: Number of participants with endometrial histology findings, e.g. benign endometrium, Malignant Neoplasm, Hyperplasia WHO 2014, no atypia or Hyperplasia WHO 2014, atypia and Endometrial Polyps.
Time Frame: Up to 2 weeks after end of treatment
Population: Participants in safety analysis set with adequate tissue were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Vilaprisan (A1) | Vilaprisan (A2) | Placebo+Vilaprisan (B1) | Vilaprisan+Placebo (B2)
Number analyzed (Participants) | 18 | 20 | 17 | 22
Participants
  Benign Endometrium | 17 | 20 | 17 | 22
  Hyperplasia WHO 2014, no atypia | 0 | 0 | 0 | 0
  Hyperplasia WHO 2014, atypia | 1 | 0 | 0 | 0
  Malignant Neoplasm | 0 | 0 | 0 | 0
  Endometrial Polyps | 1 | 1 | 1 | 0

7. Secondary Outcome: Change From Baseline of Endometrial Thickness
Description: Ultrasound examinations were performed. Endometrial thickness was measured in the medio-sagittal section as double-layer in millimeters. Summary statistics for change from baseline in endometrial thickness was provided in below table.
Time Frame: Treatment phase (up to 2 weeks after end of treatment) and follow-up phase (starts on the day after the end of the treatment until the last study visit [up to approximately 2 years])
Population: Participants in SAF with endometrial thickness measured and analyzed.
Measure: Mean (Standard Deviation); unit: Millimeters
Arm/Group | Vilaprisan (A1) | Vilaprisan (A2) | Placebo+Vilaprisan (B1) | Vilaprisan+Placebo (B2)
Number analyzed (Participants) | 18 | 20 | 17 | 22
Millimeters
  Treatment phase | -2.2 (3.0) | -1.3 (4.3) | -1.8 (4.9) | -1.8 (3.4)
  Follow-up phase: number analyzed (Participants) | 17 | 19 | 16 | 22
  Follow-up phase | -3.0 (4.6) | -0.5 (3.8) | -3.1 (4.0) | -1.8 (3.7)

ADVERSE EVENTS:
Time Frame: For TEAEs: From the first application of study medication up to 60 calendar days after end of treatment with study medication, an average of 26 weeks. For Post-treatment AEs: All AEs that started from Day 61 after the end of treatment with study medication, up to 73 weeks.
Description: For TEAEs: participant will be counted for both treatment groups if she received different treatments (vilaprisan or placebo) in the two treatment periods. SAF population was used.
  For Post-treatment AEs: Mistakes in the administration of study drug might have affected the assignment to treatment. In general, participants who received a different study drug to the one they were randomized to, were assigned to the treatment most often received. SAF population was used.
Groups:
- Vilaprisan - Treatment Emergent AEs: Participants who received the treatment of Vilaprisan in the study - Treatment emergent AEs.
- Placebo - Treatment Emergent AEs: Participants who received placebo in the study - Treatment emergent AEs.
- Vilaprisan (A1) - Post Treatment AEs: Vilaprisan (2 mg), 2 treatment periods of 12 weeks, separated by 1 bleeding episode - Post treatment AEs.
- Vilaprisan (A2) - Post Treatment AEs: Vilaprisan (2 mg), 2 treatment periods of 12 weeks without a break - Post treatment AEs.
- Placebo+ Vilaprisan (B1) - Post Treatment AEs: Placebo, 1 treatment period of 12 weeks, and Vilaprisan (2 mg), 1 treatment period of 12 weeks, separated by 1 bleeding episode - Post treatment AEs.
- Vilaprisan+ Placebo (B2) - Post Treatment AEs: Vilaprisan (2 mg), 1 treatment period of 12 weeks, and placebo, 1 treatment period of 12 Weeks, separated by 1 bleeding episode - Post treatment AEs.
Arm/Group | Vilaprisan - Treatment Emergent AEs | Placebo - Treatment Emergent AEs | Vilaprisan (A1) - Post Treatment AEs | Vilaprisan (A2) - Post Treatment AEs | Placebo+ Vilaprisan (B1) - Post Treatment AEs | Vilaprisan+ Placebo (B2) - Post Treatment AEs
All-Cause Mortality (participants affected / at risk) | 0/69 | 0/22 | 0/18 | 0/21 | 0/17 | 0/23
Serious Adverse Events (participants affected / at risk) | 2/69 | 1/22 | 3/18 | 6/21 | 3/17 | 6/23
Other Adverse Events (participants affected / at risk) | 30/69 | 8/22 | 9/18 | 4/21 | 6/17 | 7/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vilaprisan - Treatment Emergent AEs (N=69) | Placebo - Treatment Emergent AEs (N=22) | Vilaprisan (A1) - Post Treatment AEs (N=18) | Vilaprisan (A2) - Post Treatment AEs (N=21) | Placebo+ Vilaprisan (B1) - Post Treatment AEs (N=17) | Vilaprisan+ Placebo (B2) - Post Treatment AEs (N=23)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Adrenal mass (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cystoscopy (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Renal mass (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Menometrorrhagia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Uterine haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abnormal uterine bleeding (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hysterectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Myomectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Renal lesion excision (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Salpingectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Endometrial ablation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hysterosalpingectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vilaprisan - Treatment Emergent AEs (N=69) | Placebo - Treatment Emergent AEs (N=22) | Vilaprisan (A1) - Post Treatment AEs (N=18) | Vilaprisan (A2) - Post Treatment AEs (N=21) | Placebo+ Vilaprisan (B1) - Post Treatment AEs (N=17) | Vilaprisan+ Placebo (B2) - Post Treatment AEs (N=23)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 4 (4) | 4 (4) | 2 (2) | 0 (0) | 3 (3)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cushing's syndrome (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye swelling (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 5 (7) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
Abdominal pain lower (Gastrointestinal disorders) | 4 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 9 (10) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 4 (5) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 4 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Onychomycosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyoderma (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 5 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Blood pressure increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Blood testosterone increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cortisol increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 5 (5) | 1 (1) | 1 (1) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (1)
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fibrous histiocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 9 (10) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Poor quality sleep (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Uterine polyp (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 1 (2)
Fallopian tube cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Endometrial thickening (Reproductive system and breast disorders) | 4 (6) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Heavy menstrual bleeding (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 2 (4) | 1 (1) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hot flush (Vascular disorders) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2020-02-17): https://cdn.clinicaltrials.gov/large-docs/43/NCT03400943/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-20): https://cdn.clinicaltrials.gov/large-docs/43/NCT03400943/SAP_001.pdf